CLINICAL TRIAL: NCT07288320
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Safety, and Pharmacokinetics of NBI-1117568 in Adults With Bipolar I Disorder Who Are Currently Experiencing a Manic Episode or Manic Episode With Mixed Features, With or Without Psychotic Symptoms, and Warrant Inpatient Hospitalization
Brief Title: An Assessment of Efficacy, Safety, and Pharmacokinetics of NBI-1117568 in Adults With Bipolar I Disorder With Current Mania
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NBI-1117568-BPD2036
Record Dates: First submitted 2025-12-15; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Bipolar I Disorder; Mania
Keywords: Bipolar I Disorder; Mania; NBI-1117568
MeSH Terms: conditions — Mania

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NBI-1117568 (Experimental): Participants will receive NBI-1117568.
  Interventions: Drug: NBI-1117568
- Placebo (Placebo Comparator): Participants will receive placebo matching NBI-1117568.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NBI-1117568 — Oral administration
  Arms: NBI-1117568
Drug: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
The primary objective for this study is to evaluate the efficacy of NBI-1117568 compared with placebo on improving manic symptoms in adults with bipolar I disorder who are currently experiencing an episode of mania with or without mixed features.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has a primary diagnosis of bipolar I disorder.
* The participant has had at least 1 prior documented manic episode that required treatment.
* The participant is experiencing an acute manic episode or manic episode with mixed features, with or without psychotic symptoms.

Key Exclusion Criteria:

* Any unstable or poorly controlled medical condition or chronic disease (including history of neurological, hepatic, renal, cardiovascular, gastrointestinal, pulmonary, autoimmune, or endocrine disease that may affect study participation or results), or malignancy within 90 days before the start of screening.
* Primary diagnosis is not bipolar I disorder.
* History of clozapine treatment for treatment-resistant psychosis.
* History of psychiatric hospitalization(s) for ≥30 consecutive days during the 90 days before the start of screening.

Note: Additional inclusion/exclusion criteria may apply, per protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Young Mania Rating Scale (YMRS) Total Score at Day 21 | Baseline, Day 21

SECONDARY OUTCOMES:
Change From Baseline in Clinical Global Impression - Severity Scale (CGI-S) Score at Day 21 | Baseline, Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences

IPD SHARING:
Plan to Share IPD: No